CLINICAL TRIAL: NCT02837900
Title: A Randomized, Double-blind, Placebo-controlled, Study Evaluating the Safety and Efficacy of a Second Course of Intra-articular Injections of TPX-100 in Subjects Who Previously Received TPX-100 for Patellar Osteoarthritis Involving Both Knees
Brief Title: A Study Evaluating the Safety and Efficacy of a Second Course of TPX-100 in Subjects Who Previously Received TPX-100 for Patellar Osteoarthritis Involving Both Knees
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OrthoTrophix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TPX-100-2
Record Dates: First submitted 2016-06-29; First posted 2016-07-20 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Previous LT TX knee and right placebo (Placebo Comparator): Previous left treated knee will have placebo treatment in this protocol.
  Interventions: Drug: TPX-100 200 mg 4 times weekly for 4 weeks
- Previous RT TX knee and left placebo (Placebo Comparator): Previous right treated knee will have placebo treatment in this protocol.
  Interventions: Drug: TPX-100 200 mg 4 times weekly for 4 weeks
- Both TX with Active (Active Comparator): Both knees with receive Active
  Interventions: Drug: TPX-100 200 mg 4 times weekly for 4 weeks

INTERVENTIONS:
Drug: TPX-100 200 mg 4 times weekly for 4 weeks — Ea. subject will received active TPX-100 200mg in the Left knee
  Other Names: TPX-100 100mg Left
Drug: TPX-100 200 mg 4 times weekly for 4 weeks — TPX-100 100mg Right
  Other Names: TPX-100 100mg Left

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and preliminary efficacy of a second course of TPX-100 administered by intra-articular injection to subjects with osteoarthritis of the knee who participated in study TPX-100-1.

DETAILED DESCRIPTION:
Recruit up to 70 subjects whom participated in protocol TPX-100-1. The opposing knee that was treated will be getting 200mg in 4 weekly injections. The knee that was treated in TPX-100-1 will get randomized to either 200mg dose or a placebo lookalike. The investigators will follow these subjects for 6 months. Two MRIs of bi-lateral knees will be assessed. Also collection of ADA samples at 4 time points through the 6 month period.

ELIGIBILITY:
Inclusion Criteria:

1. Previous enrollment in study TPX-100-1

   * Cruciate and collateral ligament stability as defined by clinical examination
2. Able to read, understand, sign and date the subject informed consent
3. Willingness to use only acetaminophen as the primary analgesic (pain-relieving) study medication during the injection period and through study day 30. The maximum dose of acetaminophen must not exceed 2 grams/day (2000 mg per day).
4. Willingness to use only hydrocodone or hydrocodone/acetaminophen (e.g. Norco) for breakthrough pain through study day 30.
5. Willingness not to use non-steroidal anti-inflammatory drugs (NSAIDS) such as aspirin, ibuprofen, naproxen through study day 30.
6. Female subjects of child bearing potential who are sexually active (non-abstinent) must agree to and comply with using 2 highly effective methods of birth control (oral contraceptive, implant, injectable or indwelling intrauterine device, condom with spermicide, or sexual abstinence) while participating in the study.

Exclusion Criteria:

1. "Possibly, probably or definitely" drug-related SAEs in TPX-100-1; severe or ongoing "possibly, probably or definitely" related AEs in TPX-100-1.
2. Contraindication to MRI, including: metallic fragments, clips or devices in the brain, eye, or spinal canal; implanted devices that are magnetically programmed; weight > 300 lbs.; moderate or severe claustrophobia; previous intolerance of MRI procedure
3. Prior surgery in the knees, excluding procedures for debridement only (no previous microfracture procedure)
4. Joint replacement or any other knee surgery planned in the next 12 months
5. History of rheumatoid arthritis, psoriatic arthritis, or any other autoimmune or infectious cause for arthritis
6. Knee effusion > 2+ on the following clinical scale:

   * Zero = No wave produced on downstroke
   * Trace = Small wave on medial side with downstroke
   * 1+ = Larger bulge on medial side with downstroke
   * 2+ = Effusion spontaneously returns to medial side after upstroke (no downstroke necessary)
   * 3+ = So much fluid that it is not possible to move the effusion out of the medial aspect of the knee screening
7. Last viscosupplementation (e.g. Synvisc® or similar hyaluronic acid product) injected into either knee < 3 months before screening
8. Last intra-articular knee injection of corticosteroids < 2 months before screening
9. Use of any steroids (except inhaled corticosteroids for respiratory problems) during the previous month before screening
10. Known hypersensitivity to TPX-100
11. Known hypersensitivity to acetaminophen or hydrocodone
12. History of arthroscopy in either knee in the last 3 months before screening
13. History of septic arthritis, gout or pseudo-gout, of either knee in previous year before screening
14. Clinical signs of acute meniscal tear (locking, new acute mechanical symptoms consistent with meniscal tear)
15. Patellar chondrocalcinosis on X-Ray
16. Skin problem, rash or hypersensitivity, affecting either knee at the injection site
17. Bleeding problem, platelet or coagulation deficiency contraindicating, in the doctor's opinion, intra-articular injection
18. Active systemic infection
19. Current treatment or treatment within the previous 2 years prior to the Screening Visit for any malignancy except basal cell or squamous cell carcinoma of the skin, unless with specific written permission is provided by the Sponsor's medical monitor
20. Women of childbearing potential who are pregnant, nursing, or planning to become pregnant, and those who do not agree to remain on an acceptable method of birth control throughout the entire study period
21. Participation in other clinical osteoarthritis drug studies, with the exception of TPX-100-1, within one year prior to screening
22. Currently taking Paclitaxel (mitotic inhibitor), natalizumab (anti-integrin monoclonal antibody), or any other anti-integrin treatment.
23. History of significant liver disease or consumption of more than 3 alcoholic drinks a day. (Definition of one alcoholic drink: 12-ounces of beer, 8-ounces of malt liquor, 5-ounces of wine, 1.5-ounces or a "shot" of 80-proof distilled spirits or liquor such as gin, rum, vodka, or whiskey).

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. evaluate the safety, tolerability, and preliminary efficacy of a second course of TPX-100 who participated in study TPX-100-1 | Follow subjects for 6 months
  Safety, Tolerability and primary efficacy

SECONDARY OUTCOMES:
Change in patellar cartilage thickness in each knee as measured on standardized MRI from baseline to 6 months. | Follow subjects for 6 months
  Longitudinal changes in Patellar compartment cartilage thickness/thinness

IPD SHARING:
Plan to Share IPD: Undecided